CLINICAL TRIAL: NCT07184450
Title: Clinical Study of BCMA/CD70 Targeting Chimeric Antigen Receptor T Lymphocytes(CAR-T) in the Treatment of Refractory Pediatric Rheumatic Diseases
Brief Title: Clinical Study of BCMA/CD70-targeted CAR-T Therapy for Refractory Pediatric Rheumatic Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC103
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Juvenile Dermatomyositis (JDM); Polyarticular Juvenile Idiopathic Arthritis; Systemic Sclerosis (SSc); Primary Sjogren's Syndrome
Keywords: CAR-T; BCMA/CD70
MeSH Terms: conditions — Dermatomyositis; Arthritis, Juvenile; Scleroderma, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA/CD70-targeted CAR-T (Experimental): The experiment was divided into two phases: dose exploration (Part A) and dose extension (Part B).In Part A, three dose groups (0.3×10^5/kg, 1×10^5/kg, 3×10^5/kg) are set up, starting from the low dose group to explore the safe and effective dose.Upon the completion of Part A, 1 optimal dose is selected to enter into the Part B stage. The group will then be enrolled in 1~2 cases to continue to validate the safety and efficacy.The enrollment of 4-11 patients is expected in the each indication of the trial.
  Interventions: Biological: BCMA/CD70-targetd CAR-T

INTERVENTIONS:
Biological: BCMA/CD70-targetd CAR-T — Subjects underwent lymphocytetion cheotherapy and then received a single intravenous cell infusion

SUMMARY:
This is an investigator-initiated trial to evaluate the efficacy and safety of BCMA/CD70-targeted CAR-T in the treatment of refractory pediatric rheumatic diseases.

DETAILED DESCRIPTION:
Pediatric rheumatic diseases include juvenile dermatomyositis（JDM）, polyarticular juvenile idiopathic arthritis, systemic sclerosis（SSc）, primary Sjogren's syndrome, etc.

Juvenile dermatomyositis (JDM) is a non-suppurative chronic autoimmune disease and the most common type of juvenile idiopathic inflammatory myopathy. Its clinical manifestations include proximal limb muscle weakness and various rashes, which may be accompanied by multiple system involvement such as respiratory, cardiovascular, digestive and nervous systems.Juvenile idiopathic arthritis (JIA) is mainly characterized by chronic synovitis of the joints and also may be accompanied by functional damage to multiple organs. It is an important cause of disability and blindness in childhood. Polyarticular type is a relatively common subtype of JIA, with severe joint symptoms. Systemic sclerosis (SSc) is characterized by thickened and hardened skin and can also affect internal organs. Sjogren's syndrome (SS) is a systemic autoimmune disease that affects exocrine glands. The clinical manifestations of SS in children are mainly recurrent parotitis, parotid gland swelling and systemic symptoms.Despite the active treatment measures, these patients are still intolerant or unresponsive to the treatment, resulting in a high disability and mortality rate.

CAR-T therapy is an adoptive cell therapy that uses genetic modification technology to reprogram T cells and eliminate target cells expressing disease-related antigens through antigen-specific recognition.Since 2019, CAR-T cell therapy has been successfully applied to autoimmune diseases.Many kinds of autoimmune diseases such as systemic lupus erythematosus，systemic sclerosis, idiopathic inflammatory myopathy have good therapeutic effect. These results suggest that CAR-T cells may play a role in several different B-cell-mediated and autoantibody-driven human autoimmune diseases, which is expected to bring breakthroughs in the treatment of refractory pediatric rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥5 years old.
* To meet the diagnostic criteria of refractory B-cell-related pediatric rheumatic diseases, including but not limited to juvenile dermatomyositis, polyarticular juvenile idiopathic arthritis, systemic sclerosis, and primary Sjogren's syndrome.

  1. Diagnosed as juvenile dermatomyositis(JDM) according to the criteria of Bohan and Peter, and meeting the following conditions:

     1. The classification criteria of RJDM must meet (1) and any one of (2)-(5): (1) Patients who are intolerant or unresponsive to glucocorticoids and at least 2 immunosuppressants, and the duration of adequate hormone therapy should be at least 6 months; (2) The disease progresses rapidly and/or involves organs such as lungs, heart and gastrointestinal tract; (3) Calcification of subcutaneous or muscle and joint tissues; (4) Repeated rashes or skin ulcers; (5) Repeated or persistent myasthenia(muscle MRI indicates extensive, diffuse edema or the Childhood Myositis Assessment Scale(CMAS) should be less than 48 points, and at least two of the following five core measurement indicators should have abnormal results: Physician Global Assessment(PhGA) ≥2cm, Patient Global Assessment(PtGA) ≥2cm, Disease Activity Score(DAS) ≥2 points, Childhood Health Assessment Questionnaire(C-HAQ) ≥0.25 points, muscle enzyme level > 1.5×upper limit of normal);
     2. RJDM with anti-synthetase syndrome who are positive for anti-synthetase antibody and those with immune-mediated necrotizing myopathy who are positive for SRP or HMGCR antibody can be included.
  2. Meet the classification criteria for polyarticular juvenile idiopathic arthritis as defined by the International League of Associations for Rheumatology(ILAR) classification in 2001, and meeting the following conditions: After at least 6 months of traditional DMARDS treatment and at least one stable dose of DMARDS or biologic agent for ≥12 weeks, the disease is still active, that is, there are at least 2 active joints (defined as swollen joints; if there is no swelling, there must be limited passive range of motion, accompanied by pain during movement or joint tenderness).
  3. Meet the classification criteria for Systemic sclerosis (SSc) as defined by the 2013ACR/EULAR standards, and meeting the following conditions:

     1. Meet the definition of intractable disease: Glucocorticoids (≥0.5mg/kg/d) and cyclophosphamide, as well as one or more of the following immunomodulators (including antimalarial drugs, azathioprine,mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, beliumab, and telitacicept, etc.), did not show significant remission of the disease for more than 3 months; Or meet the criteria for rapid disease progression , clinical routine treatment is ineffective, and the benefits outweigh the risks as determined by the investigator and the patient's or guardian's full and informed consent can be considered for inclusion;
     2. Modified Rodnan Skin Score (mRSS) ≥15 points (total 51 points).
  4. Meet the classification criteria for primary Sjogren's syndrome as defined by the 2002 ACEG classification criteria /2016 EULAR/ACR classification criteria, and meeting the following conditions:

     1. Meet (1) and any one of (2)-(6): (1) For those who are intolerant or have an insufficient response to glucocorticoid (prednisone 1-2 mg/kg/d or an equivalent dose of other hormones) and at least two immunosuppressants, the duration of hormone treatment should be at least 6 months; (2) The disease progresses rapidly and/or involves organs such as the kidneys, nervous system, and lungs; (3) Repeated parotid gland swelling or repeated parotitis; (4) Recurrent rashes or skin ulcers; (5) Involvement of the blood system, repeated leukopenia, anemia or thrombocytopenia; (6) cryoglobulinemia;
     2. Positive for anti-SSA /Ro antibody;
     3. ESSDAI score ≥5 points or clinESSDAI score ≥5 points.
* Positive expression of CD19 in peripheral blood B cells determined by flow cytometry, and B cells > 5 per/uL.
* Previously not treated with CAR-T; or recurrence or poor efficacy after previous autologous or universal CD19-targeted CAR-T treatment (evaluated by the researcher).
* The functions of important organs are basically normal:

  1. Cardiac function: left ventricular ejection fraction (LVEF) ≥55%, no obvious abnormality in electrocardiogram;
  2. Renal function: eGFR≥30mL/min/1.73m2;
  3. Liver function: AST and ALT≤3.0 ULN, total bilirubin ≤2.0×ULN;
  4. Lung function: SpO2≥92%.
* Meet standards for leukapheresis or intravenous blood collection, and no other contraindications for leukapheresis.
* The subject of childbearing age has a negative urine pregnancy test result and agrees to take effective contraceptive measures during the test period until 1 year after the infusion.
* The patient or his/her guardian agrees to participate in this clinical trial and signs an informed consent indicating that he/she understands the purpose and procedure of this clinical trial and is willing to participate in the study.

Exclusion Criteria:

* Severe major organ involvement related to the primary disease, such as severe pulmonary hypertension (PHA) (mean arterial pressure > 45mmHg).
* primary immunodeficiency or severe secondary immunodeficiency that has not been corrected.
* accompanied by serious or active or uncontrollable infectious diseases, including but not limited to active tuberculosis, latent tuberculosis infection, active viral hepatitis,etc.
* Evidence of active malignant disease or diagnosis of malignant tumor(including hematological malignancies and solid tumors, except resected and cured skin basal cell carcinoma).
* Congenital heart disease or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia,etc.); Or combined with a large number of pericardial effusion, serious myocarditis, etc.;Or patients with unstable vital signs who need hypertensive drugs to maintain their blood pressure.
* suffering from other diseases that require long-term use of glucocorticoids or immunosuppressants.
* Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months before screening; Acute graft-versushost disease (GVHD) of grade 2 or above was present within 2 weeks prior to screening.
* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive.
* Had received live vaccine within 4 weeks prior to screening.
* Positive blood pregnancy test.
* Situations in which other investigators consider it inappropriate to participate in the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T in the treatment of refractory pediatric rheumatic diseases [Safety and Tolerability] | 28 days
  The incidence of adverse events after CAR-T cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) including the type, frequency and severity of adverse events.
The Total Improvement Score (TIS) of CAR-T in the treatment of refractory juvenile dermatomyositis [Effectiveness] | 6 months
  The proportion of subjects who achieved the minimal, moderate, and major clinical response of the Total Improvement Score (TIS) within 6 months after reinfusion.
Minimal disease activity, inactive disease and remission of CAR-T in the treatment of refractory polyarticular juvenile idiopathic arthritis [Effectiveness] | 6 months
  The proportion of subjects who achieved minimal disease activity, inactive disease and remission within 6 months.
Ped ACR 30/50/70/90/100 of CAR-T in the treatment of refractory polyarticular juvenile idiopathic arthritis [Effectiveness] | 6 months
  The proportion of subjects who achieved Ped ACR 30/50/70/90/100 within 6 months.
mRSS of CAR-T in the treatment of refractory systemic sclerosis [Effectiveness] | 6 months
  The changes from baseline in the modified Rodnan skin score (mRSS) within 6 months.
MDAI of CAR-T in the treatment of refractory systemic sclerosis [Effectiveness] | 6 months
  The changes from baseline in modified disease activity index (MDAI) within 6 months.
EUSTAR activity index of CAR-T in the treatment of refractory systemic sclerosis [Effectiveness] | 6 months
  The changes from baseline in EUSTAR activity index within 6 months.
CRISS of CAR-T in the treatment of refractory systemic sclerosis [Effectiveness] | 6 months
  The changes from baseline in Composite Response Index (CRISS) within 6 months.
Minimal disease activity, inactive disease and remission of CAR-T in the treatment of refractory primary Sjogren's syndrome [Effectiveness] | 6 months
  The proportion of subjects who achieved minimal disease activity, inactive disease and remission within 6 months.
The STAR response rate of CAR-T in the treatment of refractory primary Sjogren's syndrome [Effectiveness] | 6 months
  The proportion of subjects who achieved the STAR response rate within 6 months.
ESSDAI of CAR-T in the treatment of refractory primary Sjogren's syndrome [Effectiveness] | 6 months
  The changes from baseline in ESSDAI within 6 months.
clinESSDAI of CAR-T in the treatment of refractory primary Sjogren's syndrome [Effectiveness] | 6 months
  The changes from baseline in clinESSDAI within 6 months.
ESSPRI of CAR-T in the treatment of refractory primary Sjogren's syndrome [Effectiveness] | 6 months
  The changes from baseline in ESSPRI within 6 months.

SECONDARY OUTCOMES:
Cmax of BCMA/CD70 CAR-T cells [PK parameter] | 3 months
  The Peak Plasma concentration (Cmax) of amplified BCMA/CD70 CAR-T cells in peripheral blood after reinfusion.
Tmax of BCMA/CD70 CAR-T cells [PK parameter] | 3 months
  The time of amplified BCMA/CD70 CAR-T cells in peripheral blood to reach the maximum concentration (Tmax).
AUC28d/90d of BCMA/CD70 CAR-T cells [PK parameter] | 3 months
  The area under the plasma concentration versus time curve at 28 days /90 days after reinfusion (AUC28d/90d).
The clearance degree of B cells [PD parameter] | 3 months
  The clearance degree of B cells at each time point.
CAR-T-related serum cytokines [PD parameter] | 3 months
  The concentration levels of CAR-T-related serum cytokines such as IL-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China